CLINICAL TRIAL: NCT00367081
Title: Pyrimethamine Plus Sulfadiazine Versus Trimethoprim Plus Sulfamethoxazole for Treatment of Toxoplasmic Encephalitis in AIDS Patients: A Randomized Controlled Trial.
Brief Title: Treatment of Cerebral Toxoplasmosis in HIV/AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVH-CTR_001
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Toxoplasmic Encephalitis; AIDS
Keywords: Toxoplasmic Encephalitis; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Pyrimethamine; Sulfadiazine

INTERVENTIONS:
Drug: TMX-SMX (Bactrim(R))
Drug: Pyrimethamine plus Sulfadiazine plus leucoverin

SUMMARY:
Neurological manifestations of Cerebral toxoplasmosis or Toxoplasmic encephalitis (TE) in most advance stage HIV infected patients composed of fever, headache, alteration of consciousness with focal neurological signs/symptoms such as include hemiparesis, cranial nerve palsies, and ataxia. Generalised convulsions, in ¾ of patients. Moreover meningeal irritation sign or herniation sign may be presented as life threatening condition

DETAILED DESCRIPTION:
Background: Toxoplasmic encephalitis (TE), caused by Toxoplasma gondii, is common in AIDS patients. TE can result in tissue destruction via massive inflammation and brain abscess formation. METHODS: Randomized controlled trials were performed in AIDS patients to assess which drug regimen was optimally effective for the treatment of TE. AIDS patients with TE were randomly divided into 3 groups that received a 6-week course of either pyrimethamine (50 mg/ day or 100 mg/day) plus sulfadiazine (4 g/day) and folinic acid (25 mg/day) or trimethoprim (10 mg/kg/day) plus sulfamethoxazole (50 mg/kg/day) (TMP-SMX), and results were evaluated with respect to clinical response, mortality, morbidity, and serious adverse events. The primary outcome was defined as death in the first 6-week period. The secondary outcome was successful treatment within 6 weeks without severe adverse events, bone marrow suppression, drug-induced rash, or any other event that caused a change in the treatment regimen. RESULTS: The results from this study showed that in AIDS patients, TE was most successfully treated with the combination of pyrimethamine (50 mg/day) plus sulfadiazidine (4 g/day) and folinic acid (25 mg/day); failure rates were not significantly different among the 3 treatment groups. Conclusions: Available data suggest that of the currently available options, treatment of TE with pyrimethamine at 50 mg/day plus sulfadiazidine at 4 g/day provides the best primary outcome for AIDS patients with TE; however, because this study was terminated prematurely, we suggest that treatment with intravenous TMP-SMX be further evaluated to determine its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* AIDS
* Age > 16 years
* Clinical Diagnosis of Cerebral toxoplasmosis, Toxoplasmic encephalitis
* Positive serum titer for Toxoplasma gondii or Positive CSF titer for Toxoplasma gondii after treatment within 2 weeks
* CT scan suspected toxoplasmosis, ring enhancing lesion
* CD4<200

Exclusion Criteria:

* Sulfa drugs allergy
* positive lymphoma cell cytology in CSF
* no informed consent by patients or first degreee relatives
* CD4 >200

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-05; Study Completion 2004-08

PRIMARY OUTCOMES:
Survival rate

SECONDARY OUTCOMES:
Complete medication rate

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Chiang Mai University hospital (2003-2004), Chiang Mai, Thailand

REFERENCES:
- [Result] Kongsaengdao S, Samintarapanya K, Oranratnachai K, Prapakarn W, Apichartpiyakul C. Randomized controlled trial of pyrimethamine plus sulfadiazine versus trimethoprim plus sulfamethoxazole for treatment of toxoplasmic encephalitis in AIDS patients. J Int Assoc Physicians AIDS Care (Chic). 2008 Jan-Feb;7(1):11-6. doi: 10.1177/1545109707301244. Epub 2007 May 21. PMID 17517949